CLINICAL TRIAL: NCT05653648
Title: Testing the Feasibility of Resistant Starch From Potatoes to Modify Short-chain Fatty Acid Levels After Bariatric Surgery
Brief Title: Fiber Supplementation After Bariatric Surgery
Acronym: FSPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer L. Meijer, Assistant Professor, Department of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Study02001775
Record Dates: First submitted 2022-12-06; First posted 2022-12-16 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Potato Starch Supplement (Experimental): Participants will consume a 24 grams of potato starch on Days 1-15 and 48 grams of potato starch on Days 16-30.
  Interventions: Dietary Supplement: Potato starch

INTERVENTIONS:
Dietary Supplement: Potato starch — Participants will consume 24 grams (days 1-15) and 48 grams (days 16-30) of potato starch. Potato starch is a type 2 resistant starch that is available over the counter.

SUMMARY:
Test compliance and gastrointestinal tolerance of a 30-day dose of potato starch in bariatric patients, and determine if short chain fatty acids, specifically butyrate, increase in response to the dosages of potato starch.

DETAILED DESCRIPTION:
Despite the successful weight loss associated with bariatric surgery, epidemiology studies have observed conflicting associations between bariatric surgery and incidence of colorectal cancer (CRC), potentially suggesting an increased risk of CRC post-surgery. The investigators have identified a potential mechanism between bariatric surgery and CRC via profiling dietary intake, gut microbiota colonization, and short-chain fatty acid (SCFA) production, including acetate, propionate, and butyrate. They have demonstrated a decrease in SCFA after bariatric surgery. As intestinal SCFAs inhibit colon cancer cell proliferation, these results may suggest a mechanism linking bariatric surgery, SCFA levels, and CRC.

The objective of this protocol is to implement a 30-day fiber supplement, made from potato starch, as previous studies have successfully demonstrated that a resistant starch supplement increases intestinal SCFAs in healthy populations. The resistant starch supplement will be initiated 90-days post-bariatric surgery, which is when fiber supplements are tolerated. Fecal samples will be collected pre- and post-supplement and a targeted liquid chromatography/mass spectrometry platform will quantify levels of SCFAs. As SCFA levels have been associated with reduced hunger in other studies, the investigators will determine if hunger levels are altered in response to the supplement. The proposed study is described in the following aims:

Specific Aim 1. Assess compliance and gastrointestinal tolerance of a 30-day dose of potato starch in bariatric patients.

Specific Aim 2. Determine if short chain fatty acids, specifically butyrate, increase in response to the dosages of potato starch.

Exploratory Aim. Determine if there are changes in dietary intake, appetite, and satiety in response to the dosages of potato starch.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* Bariatric surgery at Dartmouth Medical Center
* Daily protein intake ≥ 60 grams
* Daily fluid intake ≥ 48 fl oz.

Exclusion Criteria:

* > 550 lbs at bariatric surgery date.
* Allergies to potato starches.
* Surgical complications per bariatric team members
* Individuals who cannot speak and/or write in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | 30 days
  Test gastrointestinal tolerance of a 30-day dose of potato starch in bariatric patients. Gastrointestinal tolerance will be measured using the GSRS survey (Svedlund et al, Digestive Diseases and Sciences, 1988). Statistics will use paired t-test.

SECONDARY OUTCOMES:
Short-chain fatty acid | 30 days
  Test changes in short-chain fatty acid levels from stool samples after a 30-day dose of potato starch in bariatric patients. Statistics will use paired t-test.

OTHER OUTCOMES:
Hunger and food cravings | 30 days
  Test hunger and food craving changes after a 30-day dose of potato starch in bariatric patients. Hunger and food cravings will be measured using the Control of Eating Questionnaire survey (Dalton et al, EJCN, 2015). Statistics will use paired t-test.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
Metabolomics data will be uploaded to Metabolomics Workbench one year after receiving data. Clinical variables, dietary data, and survey responses will be available upon request to PI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available Jan 1, 2024 - indefinitely.